CLINICAL TRIAL: NCT05090826
Title: A Real-World Study Evaluating Clinical Outcomes in China for the TECNIS Synergy™ Intraocular Lens Model ZFR00V
Brief Title: A Real-World Study for the TECNIS Synergy™ Intraocular Lens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Surgical Vision, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PCOL-201-CHSN
Record Dates: First submitted 2021-10-12; First posted 2021-10-25 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Cataracts
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TECNIS Synergy IOL (Experimental): Model ZFR00V
  Interventions: Device: Model ZFR00V

INTERVENTIONS:
Device: Model ZFR00V — Investigational intraocular lens replaces the natural lens removed during cataract surgery in one or both eyes.

SUMMARY:
This is a prospective and retrospective, single-center, single-arm, open-label clinical study of the TECNIS Synergy™ IOL. The study will enroll up to 100 subjects from a single site in China. All implanted subjects will be followed for 12 months postoperatively.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients at least 22 years of age
2. Have/had a cataract in one or both eyes, with planned phacoemulsification with intraocular lens implantation or a history of implantation with TECNIS Synergy intraocular lens
3. Availability, willingness and sufficient cognitive awareness to understand the purpose of the examination procedures and comply with study visits
4. Voluntary participation indicated by the study informed consent form (ICF) signed by the patient or legal guardian

Exclusion Criteria:

1. Concurrent participation or participation in any other clinical study within 30 days prior to the preoperative visit
2. Planned monovision correction (one eye designated for near correction).
3. Any other systemic or ocular disease that, in the opinion of the investigator, may affect the patient's eligibility for the study, affect visual acuity or may require surgical intervention during the course of the study (e.g., macular degeneration, cystoid macular edema, diabetic retinopathy, etc.).

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2021-12-28 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
mean monocular postoperative DCNVA | 6 months
percentage of eyes that achieve 0.3 ,0.2, 0.1 and 0.0 logMAR monocular DCNVA | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Surgical Vision Clinical Trials, Study Director — Johnson & Johnson Surgical Vision
Locations (1):
- Hainan Eye Optometry Eye Hospital Co., Ltd. No. 6, Qionghai, Hainan, China

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Medical Devices Companies have an agreement with the Yale Open Data Access (YODA) Project to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA project site at http://yoda.yale.edu
URL: http://yoda.yale.edu